CLINICAL TRIAL: NCT07074730
Title: General Anesthesia Versus Spinal Anesthesia With Local Anesthetic Infiltration for Buccal Mucosal Graft in Urethroplasty: A Randomized Controlled Trial
Brief Title: General Anesthesia Versus Spinal Anesthesia With Local Anesthetic Infiltration for Buccal Mucosal Graft in Urethroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Allah Hamdy Elbahy, Assistant lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36265MD360/1/25
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: General Anesthesia; Spinal Anesthesia; Local Anesthetic Infiltration; Buccal Mucosal Graft; Urethroplasty
MeSH Terms: interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): Spinal anesthesia with local anesthetic infiltration.
  Interventions: Other: Spinal anesthesia
- Group G (Active Comparator): General anesthesia.
  Interventions: Other: General anesthesia

INTERVENTIONS:
Other: Spinal anesthesia — Patients will receive spinal anesthesia with local anesthetic infiltration.
  Arms: Group S
Other: General anesthesia — Patients will receive general anesthesia.
  Arms: Group G

SUMMARY:
This study aims to compare general anesthesia and spinal anesthesia with local anesthetic infiltration for buccal mucosal graft (BMG) in urethroplasty.

DETAILED DESCRIPTION:
Urethroplasty is a surgical procedure aimed at reconstructing the urethra and is considered the standard treatment for bulbar urethral strictures, with different types of tissues used as either grafts or flaps, affecting approximately 300 per 100,000 males.

Postoperative pain following urethroplasty with buccal mucosal graft (BMG) is primarily related to the oral graft harvest site.

General Anesthesia provides a state of complete unconsciousness, ensuring that patients are free from pain and awareness during the surgery. It can be beneficial in complex cases or when extended manipulation is required, allowing for muscle relaxation and controlled ventilation.

On the other hand, spinal anesthesia involves the injection of anesthesia into the cerebrospinal fluid, resulting in targeted numbness in the lower body. This technique can be advantageous for its fast, simple, cost-effective method, rapid onset, lower risk of systemic complications, and preservation of airway reflexes.

ELIGIBILITY:
Inclusion Criteria:

* Male patient age ≥ 21 years.
* American Society of Anesthesiologists (ASA) classification I-II.
* Patient scheduled for urethroplasty.

Exclusion Criteria:

* Patients who are taking analgesics for chronic illness or have a history of substance abuse.
* Patients who are unable to describe their postoperative pain (e.g., neuropsychiatric disorder).
* Patients with known local anesthetics and opioid allergy.
* Patients with infection at the site of the needle puncture.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males scheduled for urethroplasty
Enrollment: 100 (Estimated)
Dates: Start 2025-07-19 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Numerical rating Scale (NRS). NRS (0 represents "no pain"; (1-3) mild pain; (4-6) moderate pain; (7-10) severe pain. NRS will be assessed at 0, 4, 8, 12, 18 and 24h postoperatively.

SECONDARY OUTCOMES:
Postoperative morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the Numerical rating Scale (NRS)> 3 to be repeated after 30 min if pain persists until the NRS< 4.
Operative time | Till discharge to post-anesthesia care unit (Up to 2 hours)
  Operative time will be recorded from the induction of anesthesia to discharge to the post-anesthesia care unit (PACU).
Length of hospital stay | Till discharge from hospital (Up to one week).
  Length of hospital stay will be recorded from admission till the discharge from the hospital.
Patient satisfaction | 24 hours postoperatively
  • Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely unsatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
Incidence of complications | 24 hours postoperatively
  Incidence of complications such as urinary retention, nausea, headache, local anesthetic systemic toxicity (LAST), bradycardia, hypotension, nausea, vomiting, respiratory depression or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.